CLINICAL TRIAL: NCT00986258
Title: An Evaluation of the Effectiveness and Tolerability of Tapentadol Hydrochloride Prolonged Release, and Tapentadol Hydrochloride Immediate Release on Demand, in Subjects With Severe Chronic Nociceptive, Mixed or Neuropathic Low Back Pain Taking WHO Step III Analgesics But Showing a Lack of Tolerability
Brief Title: Evaluation of Effectiveness and Tolerability of Tapentadol Hydrochloride in Subjects With Severe Chronic Low Back Pain Taking WHO Step III Analgesics But Showing a Lack of Tolerability
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This clinical trial was terminated early, due to slow recruitment and study drug shortages.
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 835093; 2009-010428-25 (EudraCT Number); KF5503/45 (Other: Sponsor)
Record Dates: First submitted 2009-09-28; First posted 2009-09-29 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Pain; Chronic Pain; Low Back Pain; Neuropathic Pain; Nociceptive Pain
Keywords: pain assessment; tapentadol; centrally acting analgesic
MeSH Terms: conditions — Pain; Chronic Pain; Low Back Pain; Neuralgia; Nociceptive Pain | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tapentadol Prolonged Release (Experimental): Other Names:
  * Nucynta
  * Palexia
  Interventions: Drug: Tapentadol Prolonged Release

INTERVENTIONS:
Drug: Tapentadol Prolonged Release — Participants started with 50 mg, 100 mg or 150 mg tapentadol prolonged release (PR) twice daily. Opioid rotation to tapentadol was scheduled as follows:
  * if less than 100 mg morphine equivalent start with 50 mg tapentadol PR;
  * if on 101 to 160 mg morphine equivalent daily dose start with 100 mg tapentadol PR;
  * if above 161 mg morphine equivalent daily dose start with 150 mg tapentadol PR.
  Tapentadol doses were adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis). After 5 weeks, the doses of tapentadol PR were kept stable (start of Maintenance phase). The tapentadol PR formulation was administered for up to 12 weeks. Tapentadol immediate release 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes however, participants were not permitted to dose tapentadol immediate release any more when a daily dose of 500 mg tapentadol PR was reached.
  Other Names: - Nucynta; - Palexia

SUMMARY:
The main objective of the study is to evaluate the effectiveness, tolerability, and safety of tapentadol hydrochloride prolonged release in subjects suffering from severe chronic low back pain (LBP) who are taking WHO Step III analgesics and show lack of tolerability. This is a clinical effectiveness trial designed to establish a link between anticipated clinical outcomes and the clinical practice by means of selected measures of clinical and subject-reported outcome.

The trial will compare the effectiveness of previous analgesic treatment (WHO Step III) with that of tapentadol hydrochloride prolonged release treatment during defined periods of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed an Informed Consent Form indicating that they understand the purpose of and procedures required for the trial and are willing to participate in it.
* Participants are men or non-pregnant, non-lactating women. Sexually active women must be postmenopausal, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, male partner sterilization) before entry and throughout the trial. Women of childbearing potential must have a negative pregnancy test at screening.
* Participants must be appropriately communicative to verbalize and to differentiate with regard to location and intensity of the pain.
* Participants must be at least 18 years of age.
* Participants must have a diagnosis of chronic low back pain; chronic pain defined as pain lasting for at least 3 months
* If the Participant has radicular pain, this must have been present for at least 3 months and stable for the 4 weeks before enrollment.
* Participant's pain must require a strong analgesic (defined as WHO Step III) as judged by the Investigator.
* Participants must be taking a WHO Step III analgesic on a daily basis for at least 3 months prior to the Screening Visit.
* Participants must have responded to the WHO Step III analgesic, i.e., participants must have a confirmed average pain intensity score (NRS 3) of ≤5 points during the last 3 days prior to the Screening Visit.
* Participants must report opioid-related side effects as the reason to change their analgesic.
* Participants must report a rate of satisfaction with their previous analgesic regimen not exceeding "fair" on a subject satisfaction with treatment scale (5-point VRS).

Exclusion Criteria:

* Presence of a clinically significant disease or laboratory findings that in the Investigator's opinion may affect efficacy or safety assessments.
* Presence of active systemic or local infection that may, in the opinion of the Investigator, affect the efficacy, quality of life/function or safety assessments.
* History of alcohol or drug abuse, or suspicion of in Investigator's judgement.
* Presence of concomitant autoimmune inflammatory conditions.
* Known history of or laboratory values reflecting severe renal impairment.
* Known history of moderately or severely impaired hepatic function.
* History of or active hepatitis B or C within the past 3 months or history of HIV infection.
* History of seizure disorder or epilepsy.
* Any of the following within 1 year: mild/moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm. Severe traumatic brain injury within 15 years (consisting of 1 or more of the following: brain contusion, intracranial hematoma, either unconsciousness or post traumatic amnesia lasting more than 24 h) or residual sequelae suggesting transient changes in consciousness.
* Pregnant or breast-feeding.
* History of allergy to, or hypersensitivity to tapentadol hydrochloride or its excipients, or contraindications related to tapentadol hydrochloride including:
* Subjects with acute or severe bronchial asthma or hypercapnia.
* Subjects who have or are suspected of having paralytic ileus.
* Employees of the Investigator or trial site, with direct involvement in this trial or other trials under the direction of the Investigator or trial site, as well as family members of employees of the Investigator.
* Participation in another trial concurrently or within 4 weeks prior to the Screening Visit.
* Known to or suspected of not being able to comply with the protocol and the use of the investigational medicinal product.
* Use of monoamine oxidase inhibitors within 14 days before the Screening Visit.
* Non-stable dosing of selective serotonin reuptake inhibitors within 30 days before the Screening Visit (the doses must remain stable during the trial).
* Presence of concomitant painful condition other than low back pain that could confound the subject's trial assessments or self evaluation of pain, e.g., anatomical deformities, significant skin conditions such as abscess or syndromes with widespread pain such as fibromyalgia.
* Any painful procedures during the trial (e.g., major surgery) that may, in the opinion of the Investigator, affect the efficacy or safety assessments.
* Pending litigation due to chronic pain or disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2009-10-30 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schäfer, Prof. MD, Principal Investigator — Charité University Berlin, Campus Virchow Klinikum
Locations (27):
- Belgium (4):
  - BE004, Bruges
  - BE003, Charleroi
  - BE002, Edegem
  - BE001, Liège
- CZ001, Brno, Czechia
- France (2):
  - FR004, Thionville
  - FR001, Toulouse
- Germany (7):
  - DE005, Albstadt
  - DE001, Berlin
  - DE003, Berlin
  - DE006, Kiel
  - DE004, Leipzig
  - DE008, Leipzig
  - DE007, Stuttgart
- Netherlands (4):
  - NL002, Alkmaar
  - NL004, Doetinchem
  - NL003, Eindhoven
  - NL001, Tiel
- Poland (2):
  - PL002, Krakow
  - PL001, Poznan
- Spain (5):
  - ES006, Cadiz
  - ES001, Granada
  - ES003, Málaga
  - ES004, Seville
  - ES005, Valencia
- Switzerland (2):
  - CH001, Basel
  - CH002, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site.
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials

REFERENCES:
- [Result] Galvez R, Schafer M, Hans G, Falke D, Steigerwald I. Tapentadol prolonged release versus strong opioids for severe, chronic low back pain: results of an open-label, phase 3b study. Adv Ther. 2013 Mar;30(3):229-59. doi: 10.1007/s12325-013-0015-6. Epub 2013 Mar 7. PMID 23475406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of the first participant was on the 30 October 2009 and was prematurely terminated, due to slow recruitment, on 21 January 2011 (when the last subject completed the last follow-up examination).
Pre-assignment Details: The Trial had a duration of 13 weeks. The one week Observation Period did not involve dosing with Tapentadol. For Tapentadol analyses purposes the first 6 weeks of dosing with Tapentadol are reported as one period, Titration and Optimal Dose Period. The last 6 weeks on Tapentadol are reported as the Maintenance Period.
Groups:
- Tapentadol Prolonged Release: All participants started with either 50 mg, 100 mg, or 150 mg tapentadol prolonged release (twice daily). The dose of tapentadol prolonged release was adjusted to a level that provided adequate analgesia necessary to achieve a balance between pain relief and a satisfactory level of tolerability (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol prolonged release was kept stable. Tapentadol prolonged release formulation was administered for up to 12 weeks.Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol immediate release 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes however, participants were not permitted to dose tapentadol immediate release any more when a daily dose of 500 mg tapentadol prolonged release was reached.
Period: Observation Period
Arm/Group | Tapentadol Prolonged Release
Started | 136
Completed | 125
Not Completed | 11
Not completed — Not eligible to be dosed | 11
Period: Titration and Optimal Dose Period
Arm/Group | Tapentadol Prolonged Release
Started | 125
Completed | 102
Not Completed | 23
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 3
Not completed — Non-Compliance | 1
Not completed — Other | 1
Period: Maintenance Period
Arm/Group | Tapentadol Prolonged Release
Started | 102
Completed | 93
Not Completed | 9
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Tapentadol Prolonged Release: All participants started with either 50 mg, 100 mg, or 150 mg tapentadol prolonged release (twice daily). The dose of tapentadol prolonged release was adjusted to a level that provided adequate analgesia necessary to achieve a balance between pain relief and a satisfactory level of tolerability (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol prolonged release was kept stable. Tapentadol prolonged release formulation was administered for up to 12 weeks. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol immediate release 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes however, participants were not permitted to dose tapentadol immediate release any more when a daily dose of 500 mg tapentadol prolonged release was reached.
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 49
Region of Enrollment [Number; unit: participants]
  France | 1
  Czechia | 24
  Spain | 21
  Poland | 9
  Belgium | 17
  Netherlands | 14
  Germany | 34
  Switzerland | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Responded to Treatment
Description: Participants were considered responders if they reported the same or less average pain intensity over a 3 day period (NRS-3) after 6 weeks of tapentadol prolonged release treatment compared to their previous analgesic treatment (over a 3 day period on the Numeric Rating Scale) at Week 6 compared with Week-1.
Time Frame: 6 weeks
Population: Per Protocol Set. Last Observation Carried Forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 94
participants | 76

2. Secondary Outcome: Average Pain Intensity Before the Start of Tapentadol Treatment
Description: For this pain assessment, the participant was to indicate the level of average pain experienced over the previous 3 days on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 122
units on a scale | 4.8 (0.75)

3. Secondary Outcome: Change in Average Pain Intensity After 6 Weeks of Tapentadol Prolonged Release Treatment.
Description: For this pain assessment, the participant was to indicate the level of average pain experienced over the previous 3 days on an 11-point Numerical Rating Scale(NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The value indicates the change from the baseline value on the 0 to 10 scale. A negative value indicates a reduction in pain intensity from the baseline average pain intensity.
Time Frame: Baseline; End of Week 6 (6 weeks)
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 101
units on a scale | -0.9 (1.89)

4. Secondary Outcome: Change in Average Pain Intensity After 12 Weeks of Tapentadol Prolonged Release Treatment.
Description: as for outcome 3
Time Frame: Baseline; End of Week 12 (12 weeks)
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 93
units on a scale | -1.3 (2.10)

5. Secondary Outcome: Patient Global Impression of Change
Description: In the Patient Global Impression of Change (PGIC) the participant indicates the perceived change over the treatment period. The participant is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 101
participants
  Very much improved | 5
  Much improved | 29
  Minimally improved | 47
  No change | 11
  Minimally worse | 6
  Much worse | 3
  Very much worse | 0

6. Secondary Outcome: Patient Global Impression of Change
Description: as for outcome 5
Time Frame: Baseline; End of Week 12 (12 Weeks)
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 93
participants
  Very much improved | 9
  Much improved | 34
  Minimally improved | 38
  No change | 9
  Minimally worse | 2
  Much worse | 1
  Very much worse | 0

7. Secondary Outcome: Change in the Health Survey Scores Form (SF-36)
Description: The Scores Form 36 (SF-36) includes several brief questions on 8 aspects, (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. A higher score indicates an improvement in health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state. A positive mean value indicates an improvement from baseline.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT).
  For the sub-scores "Role Emotional" and "Role Physical" there were 98 participants, for sub-scores "Physical Functioning", "Vitality" and "Mental Health" there were 99 participants, for sub-score "General Health" there were 100 participants with data available for the change of these sub-scores from baseline to visit 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 101
units on a scale
  Physical Functioning | 8.4 (18.65)
  Bodily Pain | 11.6 (20.00)
  General Health | 5.9 (15.10)
  Vitality | 9.2 (17.44)
  Social Functioning | 8.0 (24.47)
  Role Emotional | -1.4 (42.26)
  Mental Health | 5.1 (16.73)
  Role Physical | 6.9 (28.89)

8. Secondary Outcome: Change in the Health Survey Scores Form (SF-36)
Description: as for outcome 7
Time Frame: Baseline; End of Week 12 (12 Weeks)
Population: Intention to Treat (ITT).
  For the sub-scores "Role Emotional" and "Role Physical", there were only 91 participants with data available for the change of these sub-scores from baseline to visit 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 93
units on a scale
  Physical Functioning | 10.5 (19.96)
  Bodily Pain | 14.1 (22.84)
  General Health | 5.7 (14.98)
  Vitality | 12.0 (21.03)
  Social Functioning | 11.7 (27.07)
  Role Emotional | 13.9 (43.06)
  Mental Health | 9.8 (17.70)
  Role Physical | 10.7 (31.65)

9. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Sub-scores and Overall Score
Description: All participants were requested to complete the NPSI (Neuropathic Pain Symptom Inventory) questionnaire at this visit. Each participant rated their own neuropathic pain symptoms by answering ten questions relating to neuropathic symptoms on an 11-point scale 0 (not present) to 10 (worst imaginable) for each question. The higher the score for a question (sub-scale) the more bothersome the symptom is for the participant.
  Results are reported as the mean for each neuropathic symptom in the sub-scale. The mean score is reported on a scale of 0 (not present in the group) to 1 (symptom has the maximum imaginable intensity for the whole group).
Time Frame: Baseline
Population: Intention to treat (ITT).
  For the sub-scores "Overall Score" and "Pressing Pain" there were only 69 participants with data available at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 71
units on a scale
  Sub-score burning pain | 0.41 (0.284)
  Sub-score pressing pain | 0.405 (0.23)
  Sub-score paroxysmal pain | 0.422 (0.221)
  Sub-score evoked pain | 0.385 (0.216)
  Sub-score paresthesia / dysthesia | 0.424 (0.233)
  Overall score | 0.408 (0.158)

10. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Sub-scores and Overall Score
Description: All participants were requested to complete the NPSI (Neuropathic Pain Symptom Inventory) questionnaire at this visit. Each participant rated their own neuropathic pain symptoms by answering ten questions relating to neuropathic symptoms on an 11-point scale 0 (not present) to 10 (worst imaginable) for each question. The higher the score for a question (sub-scale) the more bothersome the symptom is for the participant.
  Results are reported as the mean for each neuropathic symptom in a sub-scale. The mean score is reported on a scale of 0 (not present in the group) to 1 (symptom has the maximum imaginable intensity for the whole group).
Time Frame: End of Week 6
Population: Intention to treat (ITT).
  For the sub-scores "Overall Score" and "Pressing Pain" there were only 60 participants with data available at Visit 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 61
units on a scale
  Sub-score burning pain | 0.32 (0.273)
  Sub-score pressing pain | 0.322 (0.229)
  Sub-score paroxysmal pain | 0.271 (0.231)
  Sub-score evoked pain | 0.274 (0.216)
  Sub-score paresthesia / dysthesia | 0.302 (0.21)
  Overall score | 0.297 (0.178)

11. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Sub-scores and Overall Score
Description: All participants were requested to complete the NPSI (Neuropathic Pain Symptom Inventory) questionnaire at this visit. Each participant rated their own neuropathic pain symptoms by answering ten questions relating to neuropathic symptoms on an 11-point scale 0 (not present) to 10 (worst imaginable) for each question. The higher the score for a question (sub-scale) the more bothersome the symptom is for the participant.
  Results are reported as the mean (average) for each neuropathic symptom in a sub-scale.
  The mean score is reported on a scale of 0 (not present in the group) to 1 (symptom has the maximum imaginable intensity for the whole group).
Time Frame: End of Week 12
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 56
units on a scale
  Sub-score burning pain | 0.27 (0.281)
  Sub-score pressing pain | 0.302 (0.235)
  Sub-score paroxysmal pain | 0.254 (0.255)
  Sub-score evoked pain | 0.273 (0.252)
  Sub-score paresthesia / dysthesia | 0.299 (0.239)
  Overall score | 0.280 (0.211)

12. Secondary Outcome: Mean Equipotency Ratio of Tapentadol Compared to Oxycodone
Description: Tapentadol was compared to Oxycodone with Oxycodone set to 1. The average total daily dose of Tapentadol at which a pain score equivalent or below to the pain score at the end of observation period under Oxycodone was reached was documented as the equipotent or equianalgesic dose to the total daily dose of the previously used Oxycodone.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT). 35 participants with previous oxycodone treatment.
Measure: Number; unit: Ratio
Groups:
- Tapentadol: All participants started with either 50 mg, 100 mg, or 150 mg tapentadol prolonged release (twice daily). The dose of tapentadol prolonged release was adjusted to a level that provided adequate analgesia necessary to achieve a balance between pain relief and a satisfactory level of tolerability (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol prolonged release was kept stable. Tapentadol prolonged release formulation was administered for up to 12 weeks. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol immediate release 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes however, participants were not permitted to dose tapentadol immediate release any more when a daily dose of 500 mg tapentadol prolonged release was reached.
Arm/Group | Tapentadol
Number analyzed (Participants) | 35
Ratio | 5.3

13. Secondary Outcome: Mean Equipotency Ratio of Tapentadol Compared to Buprenorphine
Description: Tapentadol was compared to Buprenorphine with Buprenorphine set to 1. The average total daily dose of Tapentadol at which a pain score equivalent or below to the pain score at the end of observation period under Buprenorphine was reached was documented as the equipotent or equianalgesic dose to the total daily dose of the previously used Buprenorphine.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT). 24 participants with previous buprenorphine treatment.
Measure: Number; unit: Ratio
Arm/Group | Tapentadol
Number analyzed (Participants) | 24
Ratio | 210.0

14. Secondary Outcome: Mean Equipotency Ratio of Tapentadol Compared to Fentanyl
Description: Tapentadol was compared to Transdermal Fentanyl with Fentanyl set to 1. The average total daily dose of Tapentadol at which a pain score equivalent or below to the pain score at the end of observation period under Transdermal Fentanyl was reached was documented as the equipotent or equianalgesic dose to the total daily dose of the previously used Fentanyl.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intent to treat (ITT). 22 participants with previous transdermal fentanyl treatment.
Measure: Number; unit: Ratio
Arm/Group | Tapentadol
Number analyzed (Participants) | 22
Ratio | 250.7

15. Secondary Outcome: Mean Equipotency Ratio of Tapentadol Compared to Morphine
Description: Tapentadol was compared to Morphine with Morphine set to 1. The average total daily dose of Tapentadol at which a pain score equivalent or below to the pain score at the end of observation period under Morphine was reached was documented as the equipotent or equianalgesic dose to the total daily dose of the previously used Morphine.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intent to treat (ITT). 14 participants with previous morphine treatment.
Measure: Number; unit: Ratio
Arm/Group | Tapentadol
Number analyzed (Participants) | 14
Ratio | 3.0

16. Secondary Outcome: Mean Equipotency Ratio of Tapentadol Compared to Hydromorphone
Description: Tapentadol was compared to Hydromorphone with Hydromorphone set to 1. The average total daily dose of Tapentadol at which a pain score equivalent or below to the pain score at the end of observation period under Hydromorphone was reached was documented as the equipotent or equianalgesic dose to the total daily dose of the previously used Hydromorphone.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT). 8 participants with previous hydromorphone treatment.
Measure: Number; unit: Ratio
Arm/Group | Tapentadol
Number analyzed (Participants) | 8
Ratio | 10.5

17. Secondary Outcome: painDETECT Assessment at Baseline
Description: The painDETECT questionnaire was used to determine the possibility of the presence of a neuropathic pain component. It is a participant completed questionnaire. A total score is calculated. Participants with a score between 0 and 12 are scored as being "negative" (no neuropathic pain component). Value between 19 and 38 as being "positive" (presence of neuropathic component)". Values from 13 to 18 are scored as being "unclear".
Time Frame: Baseline
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline painDETECT Negative Group: Subgroup of participants with a score between 0 and 12.
- Baseline painDETECT Unclear Group: Subgroup of participants with a score between 13 and 18.
- Baseline painDETECT Positive Group: Subgroup of participants with a score between 19 and 38.
Arm/Group | Baseline painDETECT Negative Group | Baseline painDETECT Unclear Group | Baseline painDETECT Positive Group
Number analyzed (Participants) | 44 | 24 | 50
units on a scale | 6.5 (3.90) | 14.7 (2.39) | 21.1 (3.39)

18. Secondary Outcome: painDETECT Assessment for Participants After 6 Weeks of Tapentadol Prolonged Release Treatment
Description: The baseline painDETECT score was reassessed at the end of Week 6.
  It is a participant completed questionnaire. A total score is calculated. Participants with a score between 0 and 12 are scored as being "negative" (no neuropathic pain component). Value between 19 and 38 as being "positive" (presence of neuropathic component)". Values from 13 to 18 are scored as being "unclear".
Time Frame: End of Week 6
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline painDETECT Negative Group: The subgroup of participants scoring 0-12 at the baseline painDETECT assessment were reassessed at the end of Week 6.
- Baseline painDETECT Unclear Group: The subgroup of participants scoring 13-18 at the baseline painDETECT assessment were reassessed at the end of Week 6.
- Baseline painDETECT Positive Group: The subgroup of participants scoring 19-38 at the baseline painDETECT assessment were reassessed at the end of Week 6.
Arm/Group | Baseline painDETECT Negative Group | Baseline painDETECT Unclear Group | Baseline painDETECT Positive Group
Number analyzed (Participants) | 35 | 20 | 45
units on a scale | 7.5 (4.18) | 10.5 (4.75) | 17.4 (5.95)

19. Secondary Outcome: painDETECT Assessment for Participants After 12 Weeks of Tapentadol Prolonged Release Treatment
Description: The baseline painDETECT score was reassessed at the end of Week 12.
  It is a participant completed questionnaire. A total score is calculated. Participants with a score between 0 and 12 are scored as being "negative" (no neuropathic pain component). Value between 19 and 38 as being "positive" (presence of neuropathic component)". Values from 13 to 18 are scored as being "unclear".
Time Frame: End of Week 12
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline painDETECT Negative Group: The subgroup of participants scoring 0-12 at the baseline painDETECT assessment were reassessed at the end of Week 12.
- Baseline painDETECT Unclear Group: The subgroup of participants scoring 13-18 at the baseline painDETECT assessment were reassessed at the end of Week 12.
- Baseline painDETECT Positive Group: The subgroup of participants scoring 19-38 at the baseline painDETECT assessment were reassessed at the end of Week 12.
Arm/Group | Baseline painDETECT Negative Group | Baseline painDETECT Unclear Group | Baseline painDETECT Positive Group
Number analyzed (Participants) | 33 | 19 | 40
units on a scale | 6.8 (4.85) | 8.6 (5.43) | 16.5 (7.17)

ADVERSE EVENTS:
Time Frame: In total, subjects were to be treated for up to 12 weeks with tapentadol.
Groups:
- Tapentadol Prolonged Release: All participants started with either 50 mg, 100 mg, or 150 mg tapentadol prolonged release (twice daily). The dose of tapentadol prolonged release was adjusted to a level that provided adequate analgesia necessary to achieve a balance between pain relief and a satisfactory level of tolerability (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol prolonged release was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol immediate release 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes however, participants were not permitted to dose tapentadol immediate release once 500 mg tapentadol prolonged release dose was reached.
Arm/Group | Tapentadol Prolonged Release
Serious Adverse Events (participants affected / at risk) | 11/125
Other Adverse Events (participants affected / at risk) | 85/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Prolonged Release (N=125)
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Trachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 2
Oedema (General disorders) | 1
pneumonia (Infections and infestations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Prolonged Release (N=125)
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 13
Dry mouth (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 19
Drug Withdrawal Syndrome (General disorders) | 26
Fatigue (General disorders) | 13
Dizziness (Nervous system disorders) | 16
Headache (Nervous system disorders) | 18
Insomnia (Psychiatric disorders) | 16
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10

LIMITATIONS AND CAVEATS:
The results of this trial have to be interpreted under the consideration that it was an open-label trial which was prematurely terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Grünenthal reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.